CLINICAL TRIAL: NCT01385514
Title: Evaluating Strategies to Prevent Staphylococcus Aureus Skin and Soft Tissue Infections in Soldiers During Infantry Training
Brief Title: Staphylococcus Aureus Skin and Soft Tissue Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Other Study IDs: 1042-2011
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Staphylococcus Aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasal swabs to detect Staphylococcus aureus skin infection to detect Staphylococcus aureus
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- company A-Training Base No.1
- company A-Training Base No.2
- company A-Training Base No.3

SUMMARY:
The purpose of this study is to evaluate strategies to prevent Staphylococcus aureus skin and soft tissue infections in soldiers during infantry training.

This study will be conducted on three different bases among groups of male recruits to IDF training base. They will provide nasal swabs to detect Staphylococcus aureus carriage in two time points: 1. before mixing and training in confined settings, reflecting carriage acquired before entering 2. After 14-30 days. All soldiers will be under surveillance for skin infection until the end of the training program.

ELIGIBILITY:
Inclusion Criteria:

* new recruit for a combat training unit

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the population of the study will be selected from infantry training bases in the IDF
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2011-07; Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hartal, MD, Principal Investigator — International Diabetes Federation
Locations (1):
- Israeli Defense Forces, Tel Aviv, Israel